CLINICAL TRIAL: NCT03890952
Title: A Phase II Open Label, Two-armed Translational Study of Nivolumab in Combination With Bevacizumab for Recurrent Glioblastoma
Brief Title: Translational Study of Nivolumab in Combination With Bevacizumab for Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ulrik Lassen (Other)
Collaborators: Herlev Hospital (Other); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Ulrik Lassen, Head of Departmen, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CA209-9UP; 2017-003925-13 (EudraCT Number)
Record Dates: First submitted 2019-02-13; First posted 2019-03-26 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Adult Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Nivolumab; Bevacizumab; Angiogenesis Inhibitors

STUDY DESIGN:
Intervention Model Description: Two parallel arms, non-randomized, not for comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm B Nivolumab and bevacizumab (Experimental): Nivolumab and bevacizumab in patients not undergoing salvage surgery
  Interventions: Drug: Nivolumab; Drug: Bevacizumab
- Arm A Nivolumab and bevacizumab (Experimental): Nivolumab and bevacizumab in patients undergoing salvage surgery
  Interventions: Drug: Nivolumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Nivolumab — Treatment with the combination of Nivolumab and bevacizumab every 2 weeks
  Other Names: Checkpoint inhibitor
Drug: Bevacizumab — Treatment with the combination of Nivolumab and bevacizumab every 2 weeks
  Other Names: Angiogenesis inhibitor

SUMMARY:
The aim of this study is to make preliminary assessment of PD-L1 and other immune related biomarkers that might act as predictors of anti-tumor activity of Nivolumab in patients with recurrent glioblastoma

DETAILED DESCRIPTION:
The effect of Nivolumab in oncologic diseases is to modulate the immune system in order to generate and/or restore a durable anti-tumor response leading to clearance of tumor. Clinical data generated with Nivolumab monotherapy in a variety of settings support the hypothesis that blockade of the PD-1 pathway results in rejection of tumor by the host immune system. The precise mechanisms by which Nivolumab exerts its anti-tumor activity are still under investigation. To contribute to this knowledge, tumor tissue from primary operation for all patients and tumor tissue from patients in the surgical Arm A will be used for further analysis.

Targeted sequencing with next generation sequencing (NGS) and Genome-wide Associations Studies (GWAS) with the use of single nucleotide polymorphism (SNP)-arrays and micro-array for expression profiling will be performed in order to describe the profile of the tumor. At Rigshospitalet has initiated a program of NGS of patients with GBM after informed content, by obtaining fresh tissue from primary or relapse surgery. In the surgical group (Arm A) of this study NGS will be repeated after one dose of Nivolumab. This information will be used in combination with the clinical observations for each patient receiving the combination of Nivolumab and Bevacizumab and the aim is that these results could be useful towards finding prognostic and/or predictive biomarkers in GBM.

In order to study the interaction between tumor cells and the immune system investigation of intratumoral and peripheral changes in tumor-infiltration lymphocytes (TILs) will be performed. By looking at TILs and peripheral blood lymphocytes (PBLs) Surgical samples will be compared to sequencing of baseline surgical samples (before Nivolumab). The interaction of TILs and tumor cells will be assessed with in vitro functional assays of autologous tumor cell recognition. Functional patterns of antitumor CD8+ and CD4+ TILs and PBLs will be investigated, with assays combining characterization of major T cell functions and simultaneous surface staining of PD-1 after co-culture with autologous tumor cells. This may detect treatment-induced changes in the functional repertoires of CD4+ and CD8+ TILs both in the tumor microenvironment (TILs) and in the periphery (PBLs). It is expected that these analyses will reveal whether significant functional changes (defined as increased frequency of tumor-reactive T cells or as functional shifting from a monofunctional to a multifunctional profile) are induced in the whole repertoire of T cells, or whether these changes are restricted to PD-1 positive T cells.

Regarding the immune-reactivity, CD8 T cell recognition of tumor-specific-antigens (TSA), i.e. and mutation derived neoepitopes will be analyzed in enrolled patients. To analyze for immune reactivity on a personalized basis by comprising epitope-maps based on both mutation-derived neoepitopes and shared tumor antigens selected based on the individual tumor mRNA expression level.

For the prediction of mutation- and splice-variation derived epitopes, whole exome sequencing (WES) and mRNA sequencing will be conducted on tumor versus germline-control samples. Cancer-specific mutations, indels, frameshifts and splice variations will be mapped to predict T cell epitopes overlapping these regions based on the patient HLA type, using available prediction tools, netMHC. A pipeline for processing next-generation sequencing data into tumor-specific neo-epitope maps has been generated to include analyses of tumor heterogeneity and generate personalized peptide libraries for each patient and analyze for T cell recognition of personalized neoepitopes in each patient included in the study. A novel technology will tag and track multiple (>1000) antigen specific T cell specificities based on their peptide-MHC (pMHC) recognition motif through a pMHC multimer with a co-attached 'DNA barcode'. Through use of this technology T cell recognition will be assessed against large libraries of peptides in limited biological samples, such as tissue biopsies, TILs and peripheral blood mononuclear cells (PBMCs). Data will reveal to what extend mutation and splice-variant derived neoepitopes are contributing to immune recognition as a consequence of checkpoint inhibition. If these are significantly recognized, then they are likely to play a crucial role for the clinical response to checkpoint inhibition.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed GBM (including all histologic variants);
2. Age ≥ 18 years;
3. Evidence of radiological (MRI-scan) measurable recurrent progressive GBM evaluated by the Response Assessment in Neuro-Oncology (RANO) criteria;
4. In arm B measurable disease according to the RANO guidelines, within 14 days of starting treatment. Measurable disease after surgery on arm A is not required with radiographic evidence of recurrent disease after treatment with temozolomide and radiotherapy;
5. An interval of at least 4 weeks between prior radiotherapy or chemotherapy and enrolment on this protocol;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2;
7. Life expectancy, in the opinion of the investigator > 3 month;
8. Written informed consent obtained prior to any screening procedures. Patients must be willing and able to comply with the protocol and aware of the investigational nature of this study;
9. Patients must have adequate bone marrow function and organ function within 2 weeks of study treatment as defined by the following laboratory criteria;

   1. Hematopoietic function: total white blood cell count (WBC) ≥ 3000/mm³, absolute neutrophil count (ANC) ≥ 1500/mm³, platelet count ≥ 125,000/mm³; hemoglobin ≥ 9g/dL
   2. Hepatic function: bilirubin < 1.5 times the upper limit of normal (ULN) (excluding Gilberts Syndrome, for which bilirubin must be < 4 times ULN), ALAT < 2.5 times ULN;
   3. Renal function: serum creatinine < 1.5 ULN or estimated creatinine clearance of ≥ 50 mL/min, calculated using the formula of Cockcroft and Gault;
   4. APTT and INR < normal limit
10. All female patients and partners of childbearing potential must agree to use adequate birth control during study treatment and for 5 months after the last dose of study drug and have a negative serum pregnancy test at screening. Acceptable methods of contraception are oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, or a sexual partner who is surgically sterilized or post-menopausal.
11. Fertile males must be willing to employ adequate means of contraception during study treatment and for 7 months after the last dose of study drug;
12. Archived paraffin-embedded tissue (approximately 10 unstained slides or a tumor block) must be available for confirmation of tumor diagnosis and correlative studies;
13. Patients in the surgical arm (Arm A) must be predicted pre-operatively to have sufficiently sized recurrent tumor to allow for 500 mg of enhancing tumor and 300 mg of non-enhancing tumor to be resected;
14. Patients must be on a stable or decreasing dose of corticosteroids (or none) for at least 5 days prior to MRI and maximum of a dose of 20 mg prednisolone per day at enrollment of the study.

Exclusion Criteria:

1. Patients must not have significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy;
2. Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids (equivalent to max dose of 20 mg prednisolone per day) and stable for at least 5 days prior to day 1;
3. Any condition (medical, social, psychological), which would prevent adequate information and follow-up;
4. Any other active malignancy or previous malignancies within the last 5 years, except, adequately treated basal or squamous cell carcinoma of the skin, or carcinoma in situ;
5. Uncontrolled hypertension (systolic blood pressure (BP) > 150 mmHg and/or diastolic BP > 100 mmHg), unstable angina, congestive heart failure (CHF) of any New York Heart Association (NYHA) classification, serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia), history of myocardial infarction within 6 months of enrollment;
6. Clinically significant peripheral vascular disease
7. Evidence of bleeding diathesis, coagulopathy or taking ASA, NSAIDs or clopidogrel;
8. Patients with coagulation problems and medically significant bleeding in the month prior to start of treatment (e.g., peptic ulcer, epistaxis, spontaneous bleeding);
9. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 0, anticipation of need for major surgical procedure during the curse of the study;
10. Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 0;
11. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 0;
12. Known active hepatitis A, B or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen); hepatitis testing is not required;
13. Known HIV infection; HIV testing is not required;
14. Active infection requiring parenteral systemic antibiotics;
15. Administration of a live, attenuated vaccine within 4 weeks before first dose of Nivolumab prior to surgery in Arm A or Cycle 1 Day 1 (Arm A and B) or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks before first dose of Nivolumab prior to surgery in Arm A or Cycle 1 Day 1 (Arm A and B) or at any time during the study;
16. Severe infections within 4 weeks prior to Cycle 1 Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia;
17. Received oral or intravenous (IV) antibiotics within 2 weeks prior to Cycle 1 Day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible;
18. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug;
19. Dementia or altered mental status that would prohibit informed consent;
20. History of organ allograft;
21. History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegner´s granulomatosis, Sjogren´s syndrome, Bell´s palsy, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis;
22. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted;
23. Pregnant or breast-feeding women
24. Prior treatment with PD-1/PD-L1 inhibitors
25. Known hypersensitivity to any of the components of Nivolumab or Bevacizumab;
26. Investigational therapy (defined as treatment for which there is no regulatory authority; within 28 days prior to Cycle 1 Day 1;
27. Any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to Cycle 1 Day 1, with the following exceptions:

    a. Hormone-replacement therapy or oral contraceptives
28. Treatment with systemic immunosuppressive medications including, but not limited to: cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents within 2 weeks prior to Cycle 1, Day 1. The use of inhaled corticosteroids and mineralocorticoids (e.g. fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
29. Concurrent therapy with approved or investigational anticancer therapeutics;
30. Body weight significantly below ideal body weight in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Number of indels as determined using mRNA sequencing | 8 weeks
  whole exome sequencing (WES) and mRNA sequencing on tumor versus germline-control samples. We will map cancer-specific mutations, indels, frameshifts and splice variations, and predict T cell epitopes overlapping these regions based on the patient HLA type, using available prediction tools, netMHC

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  Progression-Free Survival (PFS) in both treatment Arms

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, MD, PHD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided